CLINICAL TRIAL: NCT00499577
Title: Phase I/II Combination Immunotherapy After ASCT for Advanced Myeloma to Study HTERT Vaccination Followed by Adoptive Transfer of Vaccine-Primed Autologous T Cells
Brief Title: Stem Cell Transplant, Chemotherapy, and Biological Therapy in Treating Patients With High-Risk or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland Greenebaum Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Carl H. June, University of Pennsylvania
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000552988; MSGCC-0610-GCC; UPCC-0610-GCC
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-08

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Pneumococcal Vaccines

ARMS (4):
- Group 1 (HLA-A2 positive) (Experimental): Patients receive the following peptides emulsified in incomplete Freund's adjuvant VG: I) hTERT I540 peptide; ii) hTERT R572Y peptide; iii) hTERT D988Y peptide; iv) survivin Sur1M2 peptide ; and v) CMV control peptide N495 subcutaneously (SC). Patients also receive sargramostim (GM-CSF) SC and pneumococcal conjugate vaccine intramuscularly.
  Interventions: Biological: CMV pp65 peptide; Biological: hTERT I540/R572Y/D988Y multipeptide vaccine; Biological: pneumococcal polyvalent vaccine; Biological: survivin Sur1M2 peptide vaccine
- Group 2 (Experimental): Patients receive pneumococcal conjugate vaccine intramuscularly and GM-CSF subcutaneously.
  Interventions: Biological: CMV pp65 peptide
- Second group 1 (Experimental): On days 14, 42, and 90 post-transplant, patients receive peptides and GM-CSF subcutaneously and pneumococcal conjugate vaccine intramuscularly.
  Interventions: Biological: CMV pp65 peptide; Biological: hTERT I540/R572Y/D988Y multipeptide vaccine; Biological: pneumococcal polyvalent vaccine; Biological: survivin Sur1M2 peptide vaccine
- Second group 2 (Experimental): On day 14, 42, 90 post-transplant, patients receive pneumococcal conjugate vaccine intramuscularly and GM-CSF subcutaneously.
  Interventions: Biological: CMV pp65 peptide

INTERVENTIONS:
Biological: CMV pp65 peptide — Given intramuscularly
Biological: hTERT I540/R572Y/D988Y multipeptide vaccine — Given subcutaneously
  Arms: Group 1 (HLA-A2 positive); Second group 1
Biological: pneumococcal polyvalent vaccine — Given intramuscularly
  Arms: Group 1 (HLA-A2 positive); Second group 1
Biological: survivin Sur1M2 peptide vaccine — Given subcutaneously
  Arms: Group 1 (HLA-A2 positive); Second group 1

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Thalidomide may stop the growth of cancer cells by stopping blood flow to the cancer. A stem cell transplant using stem cells from the patient may be able to replace immune cells that were destroyed by chemotherapy used to kill cancer cells. Giving an infusion of the donor's T cells after the transplant may help destroy any remaining cancer cells.

PURPOSE: This phase I/II trial is studying the side effects of stem cell transplant given together with chemotherapy and biological therapy and to see how well it works in treating patients with high-risk or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety of combination immunotherapy using activated T-cells and an hTERT/survivin multipeptide vaccine in the post-autotransplant (autologous stem cell transplantation) setting and whether it delays hematopoietic recovery or induces autoimmune events.
* To determine whether the strategy of infusing vaccine-primed T-cells early after transplant in conjunction with post-transplant booster immunizations leads to the induction of cellular immune responses to the putative tumor antigens hTERT ( the catalytic subunit of telomerase) and survivin.
* To determine if combination immunotherapy as delivered to arm I patients increases the frequency of delayed paraprotein responses between 60 days and 6 months post-transplant, sufficient to upgrade the maximal level of myeloma response, when compared to non-vaccinated (arm II) patients.

Secondary

* To determine if adoptive transfer of hTERT/survivin-primed T-cells in conjunction with multi-peptide booster immunizations generates cytotoxic T-cell responses to autologous myeloma cells in vivo.
* To evaluate myeloma clinical responses including the frequency of complete and partial responses and the 1 & 2-year event-free and overall survivals.
* To measure antibody responses to 4 of the 7 serotypes contained in the pneumococcal polyvalent vaccine as well as T-cell responses to the CRM-197 carrier protein and to a CMV peptide antigen.
* To evaluate levels of hTERT and survivin expression in patient myeloma cells.

OUTLINE: This is a multicenter study. Patients are stratified according to HLA-A2 status (positive vs negative). Patients are assigned to 1 of 2 treatment groups based on stratification.

* Immunization 1:

  * Group 1 (HLA-A2 positive): Patients receive the following peptides emulsified in incomplete Freund's adjuvant VG: I) hTERT I540 peptide; ii) hTERT R572Y peptide; iii) hTERT D988Y peptide; iv) survivin Sur1M2 peptide ; and v) CMV control peptide N495 subcutaneously (SC). Patients also receive sargramostim (GM-CSF) SC and pneumococcal conjugate vaccine (PCV) intramuscularly (IM).
  * Group 2: Patients receive PCV vaccine IM and GM-CSF SC.
* Steady-state T-cell harvesting:About 10 days (range 7-14) after immunization #1, all patients undergo a mononuclear cell apheresis procedure to collect steady-state T-cells that are cryopreserved for later expansion.
* Stem cell mobilization: After completion of the mononuclear cell apheresis procedure, all patients are offered DT-PACE chemotherapy for cytoreduction and stem cell mobilization. This regimen is as follows: dexamethasone once daily for 4 days; thalidomide once daily for 4 days; cisplatin IV continuously over 4 days (patients with serum creatinine levels ≥ 2.0 mg/dL do not receive cisplatin); doxorubicin hydrochloride IV continuously over 4 days; cyclophosphamide IV continuously over 4 days; etoposide IV continuously over 4 days. Patients also receive filgrastim (G-CSF) SC once daily starting on the day after completion of chemotherapy. An acceptable alternative for stem cell mobilization is to use cyclophosphamide IV over 12 hours or, for patients who require that outpatient stem cell mobilization procedures be performed, cyclophosphamide IV over 2 hours. The cyclophosphamide mobilization regimen should be used if the patient has already received DTPACE as part of the pre-transplant therapy.
* High-dose therapy: High-dose therapy will consist of melphalan IV over 20 minutes on day -1. Autologous stem cell infusion takes place on day 0, at least 18 hours after the administration of the high-dose melphalan. Stem cells are infused IV over 20-60 minutes. G-CSF SC should be administered beginning on day +5.
* Autologous T-cell expansion and infusion: Cryopreserved cells are expanded ex vivo for up to 12 days and prepared for infusion on day 2 post-transplant.
* Infusion of autologous T-cells: The costimulated ("activated") T-cells are infused over 20-60 minutes on day +2 of transplant.
* Immunizations 2, 3, and 4:

  * Group 1: On days 14, 42, and 90 post-transplant, patients receive peptides, PCV, and GM-CSF as in group I of immunization # 1.
  * Group 2: On day 14, 42, 90 post-transplant, patients receive PCV and GM-CSF as in group II of immunization # 1.
* Maintenance therapy: At day 180 post-transplant, after completion of post-transplant immunological assessments, patients receive low-dose thalidomide in the absence of disease progression or unacceptable toxicity.

Blood is collected at T-cell harvest and days 14, 60, 100, and 180 post-transplant. Samples are analyzed by quantitative CD3/CD4/CD8 studies, cellular immunoassays, antibody immunoassays, and gene expression.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myeloma meeting 1 of the following criteria:

  * Myeloma has relapsed, progressed, or failed to respond after at least one prior course of therapy (consisting of at least 2 treatment cycles or months of therapy)

    * Failure to respond would correspond to a reduction of less than or equal to 25% of the original, diagnostic serum or urine paraprotein measurement
  * Myeloma has responded partially to initial therapy but a complete response (immunofixation negative) has NOT developed after a minimum of 3 cycles or months of initial therapy
  * Myeloma has high-risk features as defined by the presence of one or more cytogenetic abnormalities known to confer a poor outcome even after standard autotransplants (e.g., complex karyotype [≥ 3 abnormalities], t(4;14), t(14;16), del (17) (p13.1), and/or chromosome 13 abnormalities)

    * May be enrolled even while in complete or near-complete remission
    * Extended disease-free survival after autotransplantation would be unexpected for these patients and therefore especially meaningful
* Must have measurable disease

  * Measurable disease may include quantifiable or detectable levels of serum or urine paraprotein

    * For patients with minimally secretory disease or non-secretory myeloma on study entry, serum free λ or κ light chain levels may be measured and used for disease monitoring if abnormal
    * Patients who are in complete remission at the time of proposed study entry (serum and urine immunofixation consistently negative) are not eligible unless their disease meets the criteria for high-risk disease
* No known history of myelodysplasia

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2 (unless due solely to bone pain)
* Creatinine ≤ 3.0 mg/dL and not on dialysis
* WBC ≥ 3,000/mm³
* Platelet count ≥ 100,000/mm³
* AST ≤ 2 times upper limit of normal
* Bilirubin ≤ 2.0 mg/dL (unless due to Gilbert's syndrome)
* LVEF ≥ 45%

  * A lower LVEF is permissible if a formal cardiologic evaluation reveals no evidence for clinically significant functional impairment
* FEV1, FVC, TLC, and DLCO ≥ 40% predicted

  * Patients who are unable to complete pulmonary function tests due to bone pain or fracture must have a high-resolution CT scan of the chest and must have acceptable arterial blood gases (room air PO_2 > 70 mmHg)
* Women of child-bearing potential and their spouses or partners must be willing to use adequate contraception for the duration of the active treatment phase of the study

  * Contraceptive measures must be continued as long as the patient remains on maintenance thalidomide in accordance with the STEPS program

Exclusion criteria

* Pregnant or nursing
* HIV, HTLV-1/2 seropositivity
* Known history of chronic active hepatitis or liver cirrhosis (if suspected by laboratory studies, should be confirmed by liver biopsy)
* Active hepatitis B (as defined by positive hepatitis B surface antigen)

  * Positive hepatitis C virus (HCV) antibody is NOT an exclusion
* History of severe autoimmune disease requiring steroids or other immunosuppressive treatments
* Active immune-mediated diseases including:

  * Connective tissue diseases
  * Uveitis
  * Sarcoidosis
  * Inflammatory bowel disease
  * Multiple sclerosis
* Evidence or history of other significant cardiac, hepatic, renal, ophthalmologic, psychiatric, or gastrointestinal disease that might increase the risks of participating in the study
* Active bacterial, viral or fungal infections.

PRIOR CONCURRENT THERAPY:

Inclusion criteria

* Recovered from any toxicities related to prior therapy or at least returned to their baseline level of organ function
* Patients should be off of glucocorticoids for at least 2 weeks and/or thalidomide therapy for at least 1 week prior to enrollment
* At least 2 weeks since prior steroid therapy or chemotherapy

Exclusion criteria

* Prior autotransplant or allogeneic transplant
* More than 4 distinct, prior courses of therapy for myeloma
* Also see Disease Characteristics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2006-12; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Toxicity at 21 and 28 days post-transplant
T-cell responses against the hTERT vaccine as measured by tetramer assays at 100 days post-transplant
Paraprotein levels in the blood or urine and serum free light chain analyses at 60 days and at 6 months post-transplant

SECONDARY OUTCOMES:
Cytotoxic T-cell responses against autologous myeloma cell at day 100 post-transplant via chromium-51 release or flow-based assays
Maximum clinical response
1 and 2-year event-free survival
Overall survival rates
CD4 and CD8 T-cell responses against cytomegalovirus (CMV) at days 60 and 100 post-transplantation by CFSE dye dilution assays
Composite binding antibody responses at days 60 and day 100 post-transplant by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Aaron P. Rapoport, MD, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (2):
- United States (2):
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Rapoport AP, Aqui NA, Stadtmauer EA, Vogl DT, Fang HB, Cai L, Janofsky S, Chew A, Storek J, Akpek G, Badros A, Yanovich S, Tan MT, Veloso E, Pasetti MF, Cross A, Philip S, Murphy H, Bhagat R, Zheng Z, Milliron T, Cotte J, Cannon A, Levine BL, Vonderheide RH, June CH. Combination immunotherapy using adoptive T-cell transfer and tumor antigen vaccination on the basis of hTERT and survivin after ASCT for myeloma. Blood. 2011 Jan 20;117(3):788-97. doi: 10.1182/blood-2010-08-299396. Epub 2010 Oct 28. PMID 21030558
- [Result] Stadtmauer EA, Vogl DT, Luning Prak E, Boyer J, Aqui NA, Rapoport AP, McDonald KR, Hou X, Murphy H, Bhagat R, Mangan PA, Chew A, Veloso EA, Levine BL, Vonderheide RH, Jawad AF, June CH, Sullivan KE. Transfer of influenza vaccine-primed costimulated autologous T cells after stem cell transplantation for multiple myeloma leads to reconstitution of influenza immunity: results of a randomized clinical trial. Blood. 2011 Jan 6;117(1):63-71. doi: 10.1182/blood-2010-07-296822. Epub 2010 Sep 23. PMID 20864577